CLINICAL TRIAL: NCT03244371
Title: Analysis of the Impact of HCV Treatment by Last Generation Direct Antiviral Agents (DAA) on Antiviral Immunity and HIV DNA Reservoir in Coinfected HIV-HCV Patients
Acronym: HCURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-31; 2016-A01028-43 (Other: IDRCB)
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: HIV Associated HCV
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Co infected HIV and HCV patients (Experimental)
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — 4 blood draws of 25 mls of blood will be performed at 4 differents time points (before treatment, 4 weeks later, at the end of the treatment and 6 months after the end of the treatment)

SUMMARY:
Spontaneous recovery of patients infected with HCV is related to the development of a cytotoxic immune response that is executed by specialized white blood cells, the CD8+ T cells, which develop a virus-specific response. In addition, the natural killer (NK) cells provide a first-line innate cytotoxic response, which is pivotal for the spontaneous clearing of HCV. In patients where HCV infection settles chronically, CD8+ T lymphocytes and NK cells fall into a state of anergy induced by chronic viral challenge. This anergic state is also found in the case of HIV infection and exacerbated by HIV-HCV coinfection. The first therapeutic strategies against HCV were based on a treatment with interferon alpha, which had an antiviral but also immunosuppressive effect. In fact, this therapeutic strategy was unable to help the recovery of the patient's immune system that would be expected after HCV cure. However, interferon-free therapeutic strategies combining first generation direct antiviral agents (DAA) showed a positive effect on HCV antiviral immunity, by enhancing the proliferative response of CD8+ T cells and the cytotoxic and proinflammatory responses of NK cells in HCV monoinfected patients (4, 5). Since HCV-targeted therapies based on combinations of the latest generation of DAA have nearly 100% cure rates and enable faster viral suppression over shorter treatment times, a positive impact of these regimens on antiviral immunity is plausible. This possibility would be particularly interesting in HIV-HCV co-infected patients, where reactivation of the innate antiviral immunity may contribute to immune defenses against both viruses. Moreover, it has been previously reported a moderate but significant and sustained decline of HIV-1 DNA in CD4 T cells from HIV-1/hepatitis C virus-coinfected patients receiving highly active antiretroviral therapy and treated with IFN alpha/ribavirin.

To date, the real impact on antiviral immunity of treatment as well as on HIV reservoir with the latest generation of DAA was not measured in HIV-HCV co-infected patients.

The aim of this study is to analyze the impact of the cure of hepatitis C on the HIV DNA reservoir and antiviral function of CD8+ and NK cells in a subgroup of patients receiving the latest generation DAAs for treatment of HCV infection, as part of a program for a reduction of the prevalence of chronic hepatitis C patients co-infected HIV-HCV set up within the Immuno-Hematology Service of the Sainte Marguerite Hospital (Research in routine care-Ethics committee Approval Sud- Méditerranée I ID RCB 2015-A01913-46/ Principal Investigator: Dr I Poizot-Martin).

The analysis of HIV DNA, NK and CD8+ T lymphocyte antiviral immune response prior, during and after anti-HCV treatment will need the collection of a biobank. Indeed, 25 mL peripheral blood will be collected at treatment initiation, during an interim assessment, at the end of treatment and six months post-treatment, for a total of 100 ml of additional blood collection. These analyzes will be performed by Dr C Tamalet for HIV DNA IHU-Méditerranée Infection, and the team of Prof. E Vivier, DHU- Marseille Immunopole for NK and CD8+ T lymphocyte antiviral immune response.

ELIGIBILITY:
Inclusion Criteria:

* HIV1 infected patient
* HCV positive serologie and RNA-HCV positive
* Starting an anti-HCV traitment with direct antiviral agent
* With an hepatic fibrosis score < 12,5KPa measured through elastometry or with a score < F4 from liver biopsy

Exclusion Criteria:

* HIV2 infected patients par le VIH2
* Positive for HBsAg,
* Cirrohtic patient (elastométry >12,5kPa or métavir score F4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
number of CD8+ at each time point of the treatment | 24 months
number of NK cells at each time point of the treatment | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided